CLINICAL TRIAL: NCT04119024
Title: Phase I Dose Escalation Study of Systemically Administered IL13Ra2 Chimeric Antigen Receptor (CAR) T Cells After a Nonmyeloablative Conditioning Regimen in Patients With Metastatic Melanoma and Other Solid Tumors
Brief Title: Gene Modified Immune Cells After Conditioning Regimen for the Treatment of Stage IIIC or IV Melanoma or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anusha Kalbasi (Other)
Collaborators: Melanoma Research Alliance (Other); California Institute for Regenerative Medicine (CIRM) (Other); City of Hope National Medical Center (Other); Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Anusha Kalbasi, Principal Investigator, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-77842; NCI-2019-05764 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-09-25; First posted 2019-10-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Recurrent Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm; Uveal Melanoma; Acral Melanoma; Neuroendocrine Tumors; Paraganglioma; Pheochromocytoma; Adrenocortical Carcinoma; Pancreatic Neuroendocrine Tumor; Thyroid Cancer; Breast Cancer; Lung Adenocarcinoma; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Uveal Melanoma; Neuroendocrine Tumors; Paraganglioma; Pheochromocytoma; Adrenocortical Carcinoma; Adenoma, Islet Cell; Thyroid Neoplasms; Breast Neoplasms; Adenocarcinoma of Lung; Squamous Cell Carcinoma of Head and Neck | interventions — Biopsy; Specimen Handling; Cyclophosphamide; fludarabine phosphate; Fluorodeoxyglucose F18; Interleukin-13; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (chemotherapy, IL13Ralpha2) (Experimental): Patients may receive cyclophosphamide IV over 60 minutes on days -5 to -3 and fludarabine phosphate IV over 15-30 minutes on days -5 to -2. Patients then receive IL13Ralpha2 CAR T cells IV on day 0. Patients also undergo biopsy at baseline and on study, CT, or PET and CT scan at screening and on study, magnetic resonance imaging (MRI) throughout the trial, and collection of blood samples throughout the trial. Patients with disease progression may receive a second cycle with an infusion of IL13Ralpha2 CAR T cells.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Fludeoxyglucose F-18; Biological: IL13Ralpha2-specific Hinge-optimized 4-1BB-co-stimulatory CAR/Truncated CD19-expressing Autologous TN/MEM Cells; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Fludeoxyglucose F-18 — Undergo FDG-PET/CT scan
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Biological: IL13Ralpha2-specific Hinge-optimized 4-1BB-co-stimulatory CAR/Truncated CD19-expressing Autologous TN/MEM Cells — Given IV
  Other Names: IL13 [EQ]BBzeta/truncated CD19[t]+ Naive and Memory T Cells; IL13 [EQ]BBzeta/truncated CD19[t]+ TN/MEM Cells; IL13Ra2-specific-hinge-optimized-4-1BB-CAR/truncated CD19-expressing Autologous TN/MEM Lymphocytes
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I trial studies the side effects and best dose of modified immune cells (IL13Ralpha2 CAR T cells) after a chemotherapy conditioning regimen for the treatment of patients with stage IIIC or IV melanoma or solid tumors that have spread to other places in the body (metastatic). The study agent is called IL13Ralpha2 CAR T cells. T cells are a special type of white blood cell (immune cells) that have the ability to kill tumor cells. The T cells are obtained from the patient's own blood, grown in a laboratory, and modified by adding the IL13Ralpha2 CAR gene. The IL13Ralpha2 CAR gene is inserted into T cells with a virus called a lentivirus. The lentivirus allows cells to make the IL13Ralpha2 CAR protein. This CAR has been designed to bind to a protein on the surface of tumor cells called IL13Ralpha2. This study is being done to determine the dose at which the gene-modified immune cells are safe, how long the cells stay in the body, and if the cells are able to attack the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of systemic administration of IL13Ralpha2-redirected CAR T cells, including determination of the maximum tolerated dose (MTD).

SECONDARY OBJECTIVES:

I. Clinical response. II. Determine the infiltration of IL13Ralpha2 CAR T cells into the tumor. III. Determine the persistence of IL13Ralpha2 CAR T cells in the peripheral blood.

EXPLORATORY OBJECTIVES:

I. Evaluate the induction of endogenous anti-tumor T cell responses in patients receiving IL13Ralpha2 CAR T cell therapy.

II. Assess for the occurrence of cytokine release syndrome in patients receiving IL13Ralpha2 CAR T cells by evaluating plasma cytokine levels.

OUTLINE: This is a dose-escalation study of IL13Ralpha2-specific hinge-optimized 4-1BB-co-stimulatory CAR/truncated CD19-expressing autologous TN/MEM cells (IL13Ralpha2 CAR T cells) followed by a dose-expansion study.

Patients may receive cyclophosphamide intravenously (IV) over 60 minutes on days -5 to -3 and fludarabine phosphate IV over 15-30 minutes on days -5 to -2. Patients then receive IL13Ralpha2 CAR T cells IV on day 0. Patients also undergo biopsy at baseline and on study, computed tomography (CT), or positron emission tomography (PET) and CT scan at screening and on study, magnetic resonance imaging (MRI) throughout the trial, and collection of blood samples throughout the trial. Patients with disease progression may receive a second cycle with an infusion of IL13Ralpha2 CAR T cells.

After completion of study treatment, patients are followed every 2-3 months for 2 years, every 6 months for 3 years, then every year for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy that is considered surgically incurable with either:

  * Stage IIIC melanoma including locally relapsed, satellite, in-transit lesions or bulky draining node metastasis
  * Stage IV melanoma including patients with known brain metastases
  * Other metastatic, non-central nervous system (CNS) solid tumor relapsed or refractory after all standard-of-care systemic therapies for which the patient is eligible
* Confirmed IL13Ralpha2 tumor expression by immunohistochemistry (immunohistochemical assay [IHA] H-Score >= 50 in at least 10% of the total tumor specimen and in at least two high-power fields)
* Age greater than or equal to 18 years old and less than 75 years old
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* A minimum of one measurable lesion defined as:

  * Meeting the criteria for measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST), OR
  * Skin lesion(s) selected as non-completely biopsied target lesion(s) that can be accurately measured and recorded by color photography with a ruler to document the size of the target lesion(s)
* Absolute neutrophil count (ANC) >= 1 x 10^9 cells/L (determined within 30-60 days prior to enrollment; re-evaluated within 14 days of beginning conditioning chemotherapy)
* Platelets >= 75 x 10^9/L (determined within 30-60 days prior to enrollment; re-evaluated within 14 days of beginning conditioning chemotherapy)
* Hemoglobin >= 9.5 g/dL (determined within 30-60 days prior to enrollment; re-evaluated within 14 days of beginning conditioning chemotherapy)
* Aspartate and alanine aminotransferases (AST, ALT) =< 2.5 x upper limit of normal (ULN) (determined within 30-60 days prior to enrollment; re-evaluated within 14 days of beginning conditioning chemotherapy)
* Total bilirubin =< 2 x ULN (except patients with documented Gilbert's syndrome) (determined within 30-60 days prior to enrollment; re-evaluated within 14 days of beginning conditioning chemotherapy)
* Creatinine < 2 mg/dL (or a glomerular filtration rate > 45) (determined within 30-60 days prior to enrollment; re-evaluated within 14 days of beginning conditioning chemotherapy)
* Patients with melanoma must have progressed following >= 1 line of systemic therapy, including immune checkpoint inhibitor and a BRAF inhibitor in combination with MEK inhibitor for patients with BRAF V600-activating mutation and is not considered to have an alternate treatment option with curative intent
* Must be willing and able to accept at least one leukapheresis procedure (This does not apply for patients receiving a second infusion of IL13R a2 CAR T cells as they will not undergo leukapheresis)
* Must be willing and able to provide written informed consent

Exclusion Criteria:

* Inability to purify >= 1 x 10^7 T cells from leukapheresis product (this does not apply to patients receiving a second infusion of IL13Ra2 CAR T cells as they will not undergo leukapheresis)
* Previously known hypersensitivity to any of the agents used in this study; known sensitivity to cyclophosphamide or fludarabine
* Received systemic treatment for cancer, including immunotherapy, within 14 days prior to initiation of conditioning chemotherapy administration within this protocol
* Clinically active brain metastases. Radiological documentation of absence of active brain metastases at screening is required for all patients. Prior evidence of brain metastasis successfully treated with surgery or radiation therapy will not be exclusion for participation as long as they are deemed under control at the time of study enrollment
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 2 weeks prior to enrollment; not including patients with primary or secondary adrenal insufficiency who require physiologic replacement with steroids, or patients on inhaled or topical steroids at standard doses
* Human immunodeficiency virus (HIV) seropositivity or other congenital or acquired immune deficiency state, which would increase the risk of opportunistic infections and other complications during chemotherapy-induced lymphodepletion. If there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Hepatitis B or C seropositivity with evidence of ongoing liver damage, which would increase the likelihood of hepatic toxicities from the chemotherapy conditioning regimen and supportive treatments. If there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* A Tiffeneau-Pinelli index < 70% of the predicted value. Subjects will be excluded if pulmonary function tests indicate they have insufficient pulmonary capability
* Patients will be excluded if they have a history of clinically significant electrocardiography (ECG) abnormalities, symptoms of cardiac ischemia or arrhythmias and have a left ventricular ejection fraction (LVEF) < 45% on a cardiac stress test (stress thallium, stress multigated acquisition scan (MUGA), dobutamine echocardiogram, or other stress test)
* Patients with ECG results of any conduction delays (PR interval > 200 ms, corrected QT (QTC) > 480 ms), sinus bradycardia (resting heart rate < 50 beats per minute), sinus tachycardia (HR > 120 beats per minute) will be evaluated by a cardiologist prior to starting the trial. Patients with any arrhythmias, including atrial fibrillation/atrial flutter, excessive ectopy (defined as > 20 ventricular premature complex [PVC]s per minute), ventricular tachycardia, 3rd degree heart block will be excluded from the study unless cleared by a cardiologist
* Pregnancy or breast-feeding. Female patients must be surgically sterile or be postmenopausal for two years, or must agree to use effective contraception during the period of treatment and for 6 months afterwards. All female patients with reproductive potential must have a negative pregnancy test (serum/urine) at screening and again within 14 days from starting the conditioning chemotherapy. The definition of effective contraception will be based on the judgment of the study investigators. Patients who are breastfeeding are not allowed on this study
* A concomitant active malignancy that would be considered to interfere with the assessment of the primary or secondary endpoints of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 90 days from the day of chimeric antigen receptor (CAR)-transgenic cell infusion
  Safety will be reported as incidence rates for adverse events, serious adverse events, and fatal adverse events for Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 3 or higher. Adverse events will be tabulated by treatment group and will include the number of patients for whom the event occurred, the rate of occurrence, and the severity and relationship to study drug.
Dose-limiting toxicity | Up to 28 days from the day of CAR-transgenic cell infusion

SECONDARY OUTCOMES:
Objective response rate | Up to 120 days
  Will be recorded following the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
Complete response (CR) | At day 30, 60, 120, and every 2-3 months for up to 2 years
Partial response (PR) | At day 60, 120, and every 2-3 months for up to 2 years
Progression-free survival | Time from study enrollment to the date of progressive disease first documented disease progression per RECIST v1.1 or death due to any cause by investigator assessment, whichever occurs first, assessed up to 2 years
Response for in-transit metastasis | Up to 2 years
Time to disease progression | The length of time from the date of CAR T cell infusion to the date of progressive disease first documented, death, or the start of secondary antitumor therapy, assessed up to 2 years
Overall survival | From the date of CAR T cell infusion in the clinical trial until death, whether related to the trial or not, assessed up to 2 years
Duration of overall complete response | From the time measurement criteria is met for CR until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years
Duration of overall response | From the time measurement criteria is met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years
IL13Ralpha2 CAR T cell persistence | At days 1, 7, 14, 30, 60, 90, and 120
IL13Ralpha2 CAR T Cell phenotypic monitoring | Up 2 years

OTHER OUTCOMES:
Cytokine release syndrome analysis | Up 2 years
Evaluation of an endogenous T cell anti-tumor response | Up 2 years
  The biopsies will be analyzed by hematoxylin and eosin staining (H&E), immunohistochemistry (IHC) to quantify the numbers of T lymphocytes. If sufficient quantity of tissue is available, the study investigators will attempt to monitor the phenotype of the TIL obtained from tumor biopsy samples by multicolor flow cytometry (FACS), and other immune monitoring assays.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Betof Warner, MD, PhD, Principal Investigator — Stanford University; Antoni Ribas, MD, PhD, Principal Investigator — University of California, Los Angeles; Yan Xing, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Institute, Stanford, California